CLINICAL TRIAL: NCT02816944
Title: Effectivity and Safety of Endoscopic Ultrasonography-guided Laser Ablation for Refractory Neoplasms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-004
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Refractory Neoplasms
Keywords: Endoscopic ultrasonography; Laser ablation
MeSH Terms: conditions — Neoplasms

ARMS (1):
- EUS-guided laser ablation for refractory neoplasms (Experimental)
  Interventions: Procedure: EUS-guided laser ablation for refractory neoplasms

INTERVENTIONS:
Procedure: EUS-guided laser ablation for refractory neoplasms

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of endoscopic ultrasonography (EUS) guided laser ablation liver, pancreas, and retroperitoneal tumors, the investigators used preoperative and postoperative US/CEUS/CT/MRI to assess lesions, and laboratory tests including the tumor markers to evaluate the general condition of patients. Intraoperative US/CEUS/CT would be applied to monitor ablation lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory neoplasms including small hepatocellular carcinoma adjacent to the gastrointestinal tract, pancreatic neuroendocrine tumor, retroperitoneal tumor with less than 3 cm in diameter;
* Patients with Child-Pugh A/B;
* Patients with PLT ≥ 50*10E9/L and PT ≤ 20s.

Exclusion Criteria:

* Patients with severe cardiopulmonary disease, intolerant endoscopy and anesthesia, upper gastrointestinal bleeding in shock, corrosive esophagitis and acute gastritis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
80 patients of refractory neoplasms with EUS-guided laser ablation-related effectivity as assessed by MRI | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Di Matteo F, Picconi F, Martino M, Pandolfi M, Pacella CM, Schena E, Costamagna G. Endoscopic ultrasound-guided Nd:YAG laser ablation of recurrent pancreatic neuroendocrine tumor: a promising revolution? Endoscopy. 2014;46 Suppl 1 UCTN:E380-1. doi: 10.1055/s-0034-1377376. Epub 2014 Sep 25. No abstract available. PMID 25254586
- [Result] Di Matteo F, Grasso R, Pacella CM, Martino M, Pandolfi M, Rea R, Luppi G, Silvestri S, Zardi E, Costamagna G. EUS-guided Nd:YAG laser ablation of a hepatocellular carcinoma in the caudate lobe. Gastrointest Endosc. 2011 Mar;73(3):632-6. doi: 10.1016/j.gie.2010.08.019. Epub 2010 Oct 27. No abstract available. PMID 21030019
- [Result] Di Matteo F, Martino M, Rea R, Pandolfi M, Panzera F, Stigliano E, Schena E, Saccomandi P, Silvestri S, Pacella CM, Breschi L, Perrone G, Coppola R, Costamagna G. US-guided application of Nd:YAG laser in porcine pancreatic tissue: an ex vivo study and numerical simulation. Gastrointest Endosc. 2013 Nov;78(5):750-5. doi: 10.1016/j.gie.2013.04.178. Epub 2013 May 13. PMID 23680175
- [Result] Di Matteo F, Martino M, Rea R, Pandolfi M, Rabitti C, Masselli GM, Silvestri S, Pacella CM, Papini E, Panzera F, Valeri S, Coppola R, Costamagna G. EUS-guided Nd:YAG laser ablation of normal pancreatic tissue: a pilot study in a pig model. Gastrointest Endosc. 2010 Aug;72(2):358-63. doi: 10.1016/j.gie.2010.02.027. Epub 2010 Jun 11. PMID 20541187
- [Result] Yoon WJ, Brugge WR. Endoscopic ultrasonography-guided tumor ablation. Gastrointest Endosc Clin N Am. 2012 Apr;22(2):359-69, xi. doi: 10.1016/j.giec.2012.04.017. PMID 22632957
- [Derived] Xu M, Xu D, Deng Z, Tian G, Jiang T. Long-term outcomes of endoscopic ultrasound-guided laser ablation for liver tumors in the caudate lobe: 5 years of experience. Scand J Gastroenterol. 2023 May;58(5):558-564. doi: 10.1080/00365521.2022.2148833. Epub 2022 Nov 22. PMID 36415178
- [Derived] Jiang TA, Deng Z, Tian G, Zhao QY, Wang WL. Efficacy and safety of endoscopic ultrasonography-guided interventional treatment for refractory malignant left-sided liver tumors: a case series of 26 patients. Sci Rep. 2016 Dec 13;6:36098. doi: 10.1038/srep36098. PMID 27958384